CLINICAL TRIAL: NCT02315209
Title: Multicentric Evaluation of UPP, UHS and Ultra Pro Comfort Plug for Inguinal Hernia Surgery Including Quality of Life Evaluation
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Magdeburg (Other)
Responsible Party: Principal Investigator, Dr.Andreas Koch MD, FACS, Member of the Scientific Board, University of Magdeburg
Other Study IDs: GR13-108
Record Dates: First submitted 2014-12-09; First posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Inguinal Hernia
Keywords: Inguinal Hernia, Quality of Life, Mesh
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: UHS, UPP, Comfort Plug — only Repairs with 3D Devices (UPP,UHS,Comfort Plug)

SUMMARY:
Outpatient services in Germany are less controlled by external quality assurance programs. Comprehensive outcome data for benchmarking or health-care decision-making are missing e.g. for day case surgery. A quality-of-life instrument specific to hernia repair with mesh has been recently proposed (Carolinas Comfort Scale, CCS) .This study evaluates the integration of CSS as part of a multicentre quality assurance scheme for day-case (outpatient) surgery.b.The Study Group on "Quality assurance in ambulatory hernia surgery" has developed and standardized Operation technique for 3D Implants. As a consequence, any deviation must be documented by the standard. The extension to other centers according to a standardized protocol took place (shadowing to learn the operational standards, training in documentation, Minimum quantity 30 interventions per year, etc.).

DETAILED DESCRIPTION:
* Rationale

  1. In the care of inguinal hernias exists a considerable diversity of methods. Germany is expected to experience a significant shift of service delivery from inpatient to outpatient care within the next few years. As a result of this, the need for quality-controlled procedures in the ambulatory use has emerged.
  2. A first register phase for open inguinal hernia was designed in 2010 and is now almost finished. After the evaluation of approximately 6,000 patient records, the process is considered to be extremely successful.
  3. As a central result of this first register phase can already be stated that the integration of 3D meshes in a standardized process proved to be extremely effective in open inguinal hernia. In all of the examined relevant parameters, a quality of care well above the status quo could be exhibited.
  4. This data quality is unique to the hernia care not only in Germany. In Contrast, the results also achieved considerable international attention. Hence, the working group received the Fruchaud prize for presenting the results of the American Hernia Society 2013. (see Annex, www.americanherniasociety.org)
* Objective

  a. Since this approach has proven successful in the first register phase in every respect, it is now to be continued for another two years in order to develop the basis to establish this concept as widespread (outpatient) standard. The central question will be investigated of whether the outstanding results of register phase 1 will also occur in a wide and distributed application to more centers. If this can be proved, the conditions based on worldwide unique scientific data (methodology and follow-up rates, see below) are created to establish the standard surgical procedure with central integration of 3D meshes (UPP UHS) as gold standard against the Lichtenstein method in the outpatient sector.
* Design

  1. Prospective multicenter observational study of online-based (daily updated) recording of all relevant pre-, peri-and postoperative data, including patient- as well as physician-specific follow up.
  2. Analysis of the most relevant patient-specific endpoints recurrence, pain and quality of life with a 4, 12 and 52 weeks follow-up and the use of psychometrically validated Carolina Comfort Scale (anonymous and tamper-resistant).
  3. Significant expansion of the participating centers with a special comparison of the quality of results between newly added centers and centers, that have been proven already.
  4. Duration: 01/01/2014 - 12/31/2015 with an additional one-year follow-up to 12/31/2016.

ELIGIBILITY:
Inclusion Criteria:

* Primary and recurrent inguinal Hernia
* Age>18ys
* using 3D devices

Exclusion Criteria:

- Age under 18 ys.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive Patients with inguinal Hernia, Age >18 ys., Mesh Augmentation with Ultra Pro Hernia System, Ultra pro Plug or Ultra pro comfort Plug
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | 4-12-52 weeks after surgery
  Evaluation with Carolina Comfort Scale

SECONDARY OUTCOMES:
Postoperative Complications | 4-12 weeks after surgery
  clinical examination
pain after Surgery | 4-12-52 weeks after surgery
  clinical examination, questionnaire, VAS
Recurrence | 4-12-52 weeks after surgery
  clinical examination

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Koch, MD, FACS, Principal Investigator — Institute for Quality Assurance in Operative Medicine; Ralph Lorenz, MD, Study Chair — Institute for Quality Assurance in Operative Medicine

REFERENCES:
- [Background] Heniford BT, Walters AL, Lincourt AE, Novitsky YW, Hope WW, Kercher KW. Comparison of generic versus specific quality-of-life scales for mesh hernia repairs. J Am Coll Surg. 2008 Apr;206(4):638-44. doi: 10.1016/j.jamcollsurg.2007.11.025. Epub 2008 Feb 1. PMID 18387468